CLINICAL TRIAL: NCT02205801
Title: A Randomized Control Trial Comparing Bilateral Superficial Cervical Plexus Block and Local Wound Infiltration in Thyroidectomy and Parathyroidectomy
Brief Title: Study of the Efficacy of Local Analgesia as an Adjunct to General Anesthesia in Thyroidectomy and Parathyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB14-0374
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Thyroid Neoplasms; Goiter, Nodular; Thyroid Nodule; Graves' Disease; Hyperparathyroidism
MeSH Terms: conditions — Thyroid Neoplasms; Goiter, Nodular; Thyroid Nodule; Graves Disease; Hyperparathyroidism | interventions — Saline Solution; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- superficial cervical block, active (Active Comparator): After induction of general anesthesia the surgeon will perform a bilateral superficial cervical plexus block using 0.25% Marcaine.
  Interventions: Procedure: Superficial Cervical Plexus Block; Drug: Marcaine
- local wound infiltration, placebo (Placebo Comparator): After induction of general anesthesia the surgeon will perform local wound infiltration using 0.9% Saline.
  Interventions: Procedure: Local Wound Infiltration; Drug: 0.9% saline
- local wound infiltration, active (Active Comparator): After induction of general anesthesia the surgeon will perform a local wound infiltration using 0.25% Marcaine.
  Interventions: Procedure: Local Wound Infiltration; Drug: Marcaine
- superficial cervical block, placebo (Placebo Comparator): After induction of general anesthesia the surgeon will perform a bilateral superficial cervical plexus block using 0.9% saline.
  Interventions: Procedure: Superficial Cervical Plexus Block; Drug: 0.9% saline

INTERVENTIONS:
Procedure: Superficial Cervical Plexus Block — 0.25% Marcaine is injected lateral to the sternocleidomastoid bilaterally (10mL on each side) after induction of anesthesia and prior to incision and scheduled thyroidectomy or parathyroidectomy.
  Arms: superficial cervical block, active; superficial cervical block, placebo
Procedure: Local Wound Infiltration — 0.50% Marcaine is injected at the site of incision (10mL) after induction of anesthesia and prior to incision and scheduled thyroidectomy or parathyroidectomy.
  Arms: local wound infiltration, active; local wound infiltration, placebo
Drug: 0.9% saline
  Arms: local wound infiltration, placebo; superficial cervical block, placebo
Drug: Marcaine
  Arms: local wound infiltration, active; superficial cervical block, active

SUMMARY:
We aim to study the effect of local anesthetic when used in conjunction with general anesthesia during thyroidectomy or parathyroidectomy. We hypothesize there is equivalent pain control between bilateral superficial cervical plexus block and local wound infiltration when used in conjunction with a general anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Surgical indication for parathyroidectomy or thyroidectomy

Exclusion Criteria:

* Patients < 18 years old
* Patient with history of chronic opioid use
* Patient with chronic pain syndromes
* Patient with allergy to marcaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymon Grogan, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Superficial Cervical Block, Active: After induction of general anesthesia the surgeon will perform a bilateral superficial cervical plexus block using 0.25% Marcaine.
  Superficial Cervical Plexus Block: 0.25% Marcaine is injected lateral to the sternocleidomastoid bilaterally (10mL on each side) after induction of anesthesia and prior to incision and scheduled thyroidectomy or parathyroidectomy.
  Marcaine
- Superficial Cervical Block, Placebo: After induction of general anesthesia the surgeon will perform a bilateral superficial cervical plexus block using 0.9% saline.
  Superficial Cervical Plexus Block: 0.25% Marcaine is injected lateral to the sternocleidomastoid bilaterally (10mL on each side) after induction of anesthesia and prior to incision and scheduled thyroidectomy or parathyroidectomy.
  0.9% saline
- Local Wound Infiltration, Active: After induction of general anesthesia the surgeon will perform a local wound infiltration using 0.25% Marcaine.
  Local Wound Infiltration: 0.50% Marcaine is injected at the site of incision (10mL) after induction of anesthesia and prior to incision and scheduled thyroidectomy or parathyroidectomy.
  Marcaine
- Local Wound Infiltration, Placebo: After induction of general anesthesia the surgeon will perform local wound infiltration using 0.9% Saline.
  Local Wound Infiltration: 0.50% Marcaine is injected at the site of incision (10mL) after induction of anesthesia and prior to incision and scheduled thyroidectomy or parathyroidectomy.
  0.9% saline
Period: Overall Study
Arm/Group | Superficial Cervical Block, Active | Superficial Cervical Block, Placebo | Local Wound Infiltration, Active | Local Wound Infiltration, Placebo
Started | 11 | 8 | 9 | 8
Completed | 11 | 8 | 9 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Superficial Cervical Block, Active | Superficial Cervical Block, Placebo | Local Wound Infiltration, Active | Local Wound Infiltration, Placebo | Total
Number analyzed (Participants) | 11 | 8 | 9 | 8 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (13.1) | 47.4 (15.5) | 48.2 (9.5) | 51.6 (15.3) | 49.4 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 8 | 4 | 27
  Male | 2 | 2 | 1 | 4 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 3 | 2 | 10
  White | 7 | 6 | 6 | 6 | 25
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Fentanyl Administration
Description: The total amount of Fentanyl administered during the procedure will be recorded.
Time Frame: During the procedure
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Superficial Cervical Block, Active | Superficial Cervical Block, Placebo | Local Wound Infiltration, Active | Local Wound Infiltration, Placebo
Number analyzed (Participants) | 11 | 8 | 9 | 8
mcg | 187.5 (89.2) | 185.7 (80.2) | 144.2 (65.0) | 156.3 (43.8)

2. Secondary Outcome: Post Operative Pain
Description: Pain scores will either be verbally reported to nursing and recorded or reported on a questionnaire. Back of neck pain scores range 0-10, throat pain scores range 0-9, incisional pain scores range 0-9 (zero means no pain and 9 or 10 means severe pain).
Time Frame: At four hour after operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Superficial Cervical Block, Active | Superficial Cervical Block, Placebo | Local Wound Infiltration, Active | Local Wound Infiltration, Placebo
Number analyzed (Participants) | 11 | 8 | 9 | 8
units on a scale
  Incision | 3 (2.6) | 2.8 (1.6) | 4.4 (2.9) | 2.9 (2)
  Back of neck | 1.4 (1.3) | 3.4 (3.4) | 2.3 (2.1) | 2.4 (2.0)
  Throat | 4.3 (1.6) | 5.3 (2.3) | 6.4 (1.9) | 3.9 (2.3)

3. Secondary Outcome: Post Operative Nausea Score
Description: Nausea scores will either be verbally reported to nursing and recorded or reported on a questionnaire. The scores range 0-9 (zero means no symptom and 9 means "very severe").
Time Frame: At 2 weeks after operation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Superficial Cervical Block, Active | Superficial Cervical Block, Placebo | Local Wound Infiltration, Active | Local Wound Infiltration, Placebo
Number analyzed (Participants) | 11 | 8 | 9 | 8
units on a scale
  Incision | 1.3 (0.5) | 1.0 (0) | 1.4 (1.1) | 1.4 (0.9)
  Back of neck | 1.7 (1.0) | 1.2 (0.4) | 1.3 (0.5) | 1.0 (0)
  Throat | 1.4 (0.8) | 1.0 (0) | 2.0 (1.5) | 1.2 (0.4)

4. Secondary Outcome: Total Pain Medication Utilization
Description: Total operative opioid dosages administered converted to effective mg of Hydromorphine.
Time Frame: At follow up appointment 1-2 weeks postoperatively
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Superficial Cervical Block, Active | Superficial Cervical Block, Placebo | Local Wound Infiltration, Active | Local Wound Infiltration, Placebo
Number analyzed (Participants) | 11 | 8 | 9 | 8
mg | 0.56 (0.43) | 0.71 (0.4) | 0.84 (0.47) | 0.79 (0.52)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Superficial Cervical Block, Active | Superficial Cervical Block, Placebo | Local Wound Infiltration, Active | Local Wound Infiltration, Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/8 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/8 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/11 | 0/8 | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT02205801/Prot_SAP_000.pdf